CLINICAL TRIAL: NCT02492945
Title: Safety and Effects of PDRN(Polydeoxyribonucleotide) Injection in Patient With Elbow Epicondylitis in Randomized Double-blind Active-control Comparative Study
Brief Title: Bundang Rehabilitative Impact Study of the Elbow Epicondylitis
Acronym: BundangRISEe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae-Young Lim, Safety and Effects of PDRN(polydeoxyribonucleotide) Injection in Patient with elbow epicondylitis in randomized double-blind active-control comparative study, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1411/276-004
Record Dates: First submitted 2015-06-26; First posted 2015-07-09 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-02

CONDITIONS: Lateral Epicondylitis
Keywords: Tennis elbow; Polydeoxyribonucleotides; Prolotherapy; Randomized controlled trial; Visual analogue scale; disability; ultrasonography
MeSH Terms: conditions — Tennis Elbow | interventions — Polydeoxyribonucleotides; Sodium; Glucose; Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDRN group (Experimental): They take the three times of the ultrasonography-guided injections for four weeks(0,2,4 weeks) under double-blind. PDRN group take ultrasonography-guided 3ml-Rejuvinex injection for the lesion( tear or tendinosis about extensor carpi radialis brevis, extensor digitorum communis, radial collateral ligament ) of lateral epicondylitis for 4 weeks.
  Interventions: Drug: 3ml-Rejuvinex
- Dextrose group (Active Comparator): They take the three times of the ultrasonography-guided injections for four weeks(0,2,4 weeks) under double-blind. Dextrose group as active control group takes the 3ml-15%-dextrose solution for same procedure: the lesion( tear or tendinosis about extensor carpi radialis brevis, extensor digitorum communis, radial collateral ligament ) of lateral epicondylitis for 4 weeks. This dextrose solution for common extensor tendons are used as prolotherapy.
  Interventions: Drug: 3ml-15%-dextrose solution

INTERVENTIONS:
Drug: 3ml-Rejuvinex — They take the three times of the ultrasonography-guided 3ml-Rejuvinex as a PDRN group for four weeks(0,2,4 weeks) under double-blind.
  Other Names: PDRN (Polydeoxyribonucleotide) sodium
  Arms: PDRN group
Drug: 3ml-15%-dextrose solution — They take the three times of the ultrasonography-guided 3ml-15%-dextrose solution injections as a Dextrose group for four weeks(0,2,4 weeks) under double-blind.
  Other Names: 15% dextrose and 0.2% lidocaine solution, mixed, total 3ml; as prolotherapy
  Arms: Dextrose group

SUMMARY:
This study is to assess the safety and effect of polydeoxyribonucleotide(PDRN) on the lateral epicondylitis with ultrasonography-guided injection of the PDRN or dextrose solution.

Condition: lateral epicondylitis

Intervention Drug: polydeoxyribonucleotide, PDRN Drug: dextrose solution, 15% as prolotherapy, active control

Phase 4

Study type: Interventional

Study design: Treatment, Parallel Assignment, Double Blind((Subject, intervention performer, Investigator, Outcomes Assessor), Randomized, Safety/Efficacy Study

Official Title: Safety and Effects of PDRN(polydeoxyribonucleotide) Injection in Patient with elbow epicondylitis in randomized double-blind active-control comparative study

Estimated Enrollment: 40

DETAILED DESCRIPTION:
Detailed Description:

40 patients that meet the inclusion criteria on screening test are assigned to one of two groups(PDRN group or 15% dextrose active control group) by randomization. They take the three times of the ultrasonography-guided injections for four weeks(0,2,4 weeks) under double-blind. PDRN group take ultrasonography-guided 3ml PDRN injection for the lesion( tear or tendinosis about extensor carpi radialis brevis, extensor digitorum communis, radial collateral ligament ) of lateral epicondylitis for 4 weeks. Active control group takes the 15% dextrose solution, 3ml for same procedure. The main outcome variables are measured at 0, 6 weeks and 3 months after 1st injection as starting point and compared differences from baseline to 3 month as primary end points within each group or between both group. Polydeoxyribonucleotide is verified whether it has the safety and effect on lateral epicondylitis with comparing to prolotherapy.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the study are

* provision of informed consent by patient
* adult men or women aged > 18 and < 65 years
* Patients had a clinical diagnosis of lateral epicondylitis based on local tenderness to palpation at lateral epicondyle and pain in that area elicited with active extension of the wrist in pronation and elbow extension
* History of pain >3 months and <2 years, failed each of the following conservative care modalities: relative rest, physical/occupational therapy, non-steroidal anti-inflammatorydrugs and two corticosteroid injections.
* Baseline elbow pain > 50 mm/100 mm using a visual analog scale (VAS) with resisted active extension of the wrist in pronation and elbow extension
* All affected elbows were screened with radiography and all proved to be normal, except for some calcifications of the common extensor origin.
* documented sonographic diagnosis of common extensor tendinosis was based on tendon echogenicity, loss of the normal echotexture and tendon thickening. We also performed the sonographic assessment of the extensor carpi radialis brevis, extensor digitorum communis and radial collateral ligament; tendinosis defined as ill- or well-defined focal/generalized hypoechogenic swollen tendon with loss of normal fibrillary pattern and focal tear defined as well-defined anechoic cleft

Exclusion Criteria:

* History of narcotic use for pain management > 1 mo, narcotic abuse
* History of alcoholic abuse
* any recent febrile or infectious disease
* corticosteroid injection within the past 3 months
* Signs of other causes for lateral elbow pain (posterior interosseous nerve entrapment, fracture or osteochondral lesion)
* History of carpal tunnel syndrome, cervical radiculopathy or neurologic disorder
* Other chronic widespread pain syndromes
* History of bleeding disorder, anemia
* Systemic disorders such as diabetes, rheumatoid arthritis,or hepatitis
* Intolerance/allergy to local anesthetics or injection corticosteroids
* history of vasovagal shock
* Pregnancy/lactation
* history of any malignancy (including hematologic and non hematologic malignancies)
* Hypotension, systolic BP <100mmHg, diastolic BP < 60mmHg
* Systemic disorders such as diabetes, rheumatoid arthritis, or hepatitis, nephropathy, Hypothyroidism.
* History of receiving a PDRN injection at any site
* Allergic reaction or hypersensitivity for PDRN
* Workers compensation or worker using both upper extremities, especially elbow and hand for most labor activity
* history of acute elbow trauma (<1 week)
* patients requiring antiplatelet medications for the treatment of heart attack, stroke, or other medical condition
* Previous surgery for elbow tendinosis or other disease at affected side
* Active bilateral elbow tendinosis within 4 weeks before randomization
* Tendon echogenicity, grade 0 and 4 were excluded; The degree of tendinosis is grade based on changes in tendon echotexture at sonographic assessment, Diagnostic ultrasound features for the RISEe

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visual analog scale (VAS) as lateral elbow pain at 3 months | 0, 6 and 12 weeks, 3 times
  Visual analog scale (100-mm VAS) with resisted active extension of the wrist in radial deviation, pronation and elbow extension

SECONDARY OUTCOMES:
Change from Baseline PRTEE(Patient-Rated Tennis Elbow Evaluation) at 3 months | 0, 6 and 12 weeks, 3 times
  PRTEE assesses the average pain and function of the affected arm during the preceding week. It consists of 2 parts, 1 assessing elbow pain (5 items) and 1 assessing function (10 items) using a numeric rating scale from 0 to 10, with 5 and 10 questions, respectively.
  Scores range from 0 (good quality-of- life, no pain or disability) to 100 (poor quality-of-life, extreme pain or disability).
Change from Baseline EQ-5D-5L at 3 months | 0, 6 and 12 weeks, 3 times
  EQ-5D-5L assess health-related quality of life(HRQOL) in tennis elbow patients. This is an instrument widely used to measure and evaluate general health status and describes general health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change from Baseline ASES elbow satisfaction at 3 months | 0, 6 and 12 weeks, 3 times
  ASES(American Shoulder and Elbow Surgeons) elbow is a currently among the most commonly used elbow self-report pain and disability outcome measures and have 18 item self-report questionnaire designed to measure pain and disability arising from elbow disorders. But In this trial, only one questionnaire about satisfaction is used.
Change from Baseline PPT(pressure pain threshold) at 3 months | 0, 6 and 12 weeks, 3 times
  PPT(pressure pain threshold, Kg/cm2 or lb ) is assessed by an algometry, Commander trademark. The algometry is comprised of a gauge attached to a hard rubber tip. Pressure was applied though the rubber surface area of 1 cm2 at a rate of 2 Kg/Cm2 per second.
  second. The instrument was placed perpendicular to the skin's surface at lateral epicondyle (site of maximal tenderness). The participants were asked to indicate when the pressure became painful based on this definition: "When you feel the sensation changes from pressure to the slightest pain inform us". Each measure site was tested three times with 1 minutes between each test. Their average was used for statistical analyses.
Change from Baseline Hand grip strength at 3 months | 0, 6 and 12 weeks, 3 times
  Its assessment is made by Takei digital hand grip dynamometer(unit = N ). For the actual testing procedure, pain-free grip strength measurements of the involved limb were conducted first. The subject was instructed to slowly squeeze the dynamometer and to stop the instant that changes from pressure to the slightest pain was experienced. Each measure site was tested three times with 1 minutes between each test. Their average was used for statistical analyses. Cf. pain-free maximum grip strength )
Change from Baseline Strength of wrist by isokinetic muscle performance test (IMPT) at 3 months | 0, 6 and 12 weeks, 3 times
  Isometric resistance strength( unit = N ) was tested with Primus RS (BTE, Baltimore, USA)) device. 5 times repetitive movements in wrist flexion/extension and pronation/supination are performed at both side. And average torque is calculated by obtaining the mean value of the torque signal for 5 repetition.
Change from Baseline Ultrasound features of the Common extensor tendon at 3 months | 0, 6 and 12 weeks, 3 times
  We used ACCUVIX V20 with an 5- to 13Hz broadband linear transducer ( SAMSUNG MEDICINE, Hongchun, Gangwondo). The transducer was aligned with the long axis of the radius over the common tendon origin. Diagnostic ultrasound of the common extensor tendon is first performed to evaluate the degree of tendinosis and to fully characterize tendon abnormalities. Seven ultrasound features of the Common extensor tendon are assessed as below. A. Grade of tendinosis, B. Tendon thickness, C. Radial collateral ligament(RCL) lesion, D. Tendon hyperemia (Power doppler), E. Cortical irregularity, F. Intratendinous calcification, G. Enthesophyte

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Kyung Do, Principal Investigator — Seoul National University Bundang Hospital; Jae-Young Lim, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Johnson GW, Cadwallader K, Scheffel SB, Epperly TD. Treatment of lateral epicondylitis. Am Fam Physician. 2007 Sep 15;76(6):843-8. PMID 17910298
- [Background] Price R, Sinclair H, Heinrich I, Gibson T. Local injection treatment of tennis elbow--hydrocortisone, triamcinolone and lignocaine compared. Br J Rheumatol. 1991 Feb;30(1):39-44. doi: 10.1093/rheumatology/30.1.39. PMID 1991216
- [Background] Sanchez M, Azofra J, Anitua E, Andia I, Padilla S, Santisteban J, Mujika I. Plasma rich in growth factors to treat an articular cartilage avulsion: a case report. Med Sci Sports Exerc. 2003 Oct;35(10):1648-52. doi: 10.1249/01.MSS.0000089344.44434.50. PMID 14523300
- [Background] Solveborn SA, Buch F, Mallmin H, Adalberth G. Cortisone injection with anesthetic additives for radial epicondylalgia (tennis elbow). Clin Orthop Relat Res. 1995 Jul;(316):99-105. PMID 7634730
- [Background] Maffulli N, Longo UG, Denaro V. Novel approaches for the management of tendinopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2604-13. doi: 10.2106/JBJS.I.01744. PMID 21048180
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Sanchez M, Anitua E, Azofra J, Andia I, Padilla S, Mujika I. Comparison of surgically repaired Achilles tendon tears using platelet-rich fibrin matrices. Am J Sports Med. 2007 Feb;35(2):245-51. doi: 10.1177/0363546506294078. Epub 2006 Nov 12. PMID 17099241
- [Background] Slater M, Patava J, Kingham K, Mason RS. Involvement of platelets in stimulating osteogenic activity. J Orthop Res. 1995 Sep;13(5):655-63. doi: 10.1002/jor.1100130504. PMID 7472743
- [Background] Randelli PS, Arrigoni P, Cabitza P, Volpi P, Maffulli N. Autologous platelet rich plasma for arthroscopic rotator cuff repair. A pilot study. Disabil Rehabil. 2008;30(20-22):1584-9. doi: 10.1080/09638280801906081. PMID 18608363
- [Background] Jacobson KA, Gao ZG. Adenosine receptors as therapeutic targets. Nat Rev Drug Discov. 2006 Mar;5(3):247-64. doi: 10.1038/nrd1983. PMID 16518376
- [Background] Cronstein BN. Adenosine, an endogenous anti-inflammatory agent. J Appl Physiol (1985). 1994 Jan;76(1):5-13. doi: 10.1152/jappl.1994.76.1.5. PMID 8175547
- [Background] Hasko G, Szabo C, Nemeth ZH, Kvetan V, Pastores SM, Vizi ES. Adenosine receptor agonists differentially regulate IL-10, TNF-alpha, and nitric oxide production in RAW 264.7 macrophages and in endotoxemic mice. J Immunol. 1996 Nov 15;157(10):4634-40. PMID 8906843
- [Background] Montesinos MC, Desai A, Delano D, Chen JF, Fink JS, Jacobson MA, Cronstein BN. Adenosine A2A or A3 receptors are required for inhibition of inflammation by methotrexate and its analog MX-68. Arthritis Rheum. 2003 Jan;48(1):240-7. doi: 10.1002/art.10712. PMID 12528125
- [Background] Polito F, Bitto A, Galeano M, Irrera N, Marini H, Calo M, Squadrito F, Altavilla D. Polydeoxyribonucleotide restores blood flow in an experimental model of ischemic skin flaps. J Vasc Surg. 2012 Feb;55(2):479-88. doi: 10.1016/j.jvs.2011.07.083. Epub 2011 Nov 3. PMID 22051873
- [Background] Altavilla D, Bitto A, Polito F, Marini H, Minutoli L, Di Stefano V, Irrera N, Cattarini G, Squadrito F. Polydeoxyribonucleotide (PDRN): a safe approach to induce therapeutic angiogenesis in peripheral artery occlusive disease and in diabetic foot ulcers. Cardiovasc Hematol Agents Med Chem. 2009 Oct;7(4):313-21. doi: 10.2174/187152509789541909. PMID 19860658
- [Background] Szabo C, Scott GS, Virag L, Egnaczyk G, Salzman AL, Shanley TP, Hasko G. Suppression of macrophage inflammatory protein (MIP)-1alpha production and collagen-induced arthritis by adenosine receptor agonists. Br J Pharmacol. 1998 Sep;125(2):379-87. doi: 10.1038/sj.bjp.0702040. PMID 9786512
- [Background] Carayannopoulos A, Borg-Stein J, Sokolof J, Meleger A, Rosenberg D. Prolotherapy versus corticosteroid injections for the treatment of lateral epicondylosis: a randomized controlled trial. PM R. 2011 Aug;3(8):706-15. doi: 10.1016/j.pmrj.2011.05.011. PMID 21871414
- [Background] Chiavaras MM, Jacobson JA, Carlos R, Maida E, Bentley T, Simunovic N, Swinton M, Bhandari M. IMpact of Platelet Rich plasma OVer alternative therapies in patients with lateral Epicondylitis (IMPROVE): protocol for a multicenter randomized controlled study: a multicenter, randomized trial comparing autologous platelet-rich plasma, autologous whole blood, dry needle tendon fenestration, and physical therapy exercises alone on pain and quality of life in patients with lateral epicondylitis. Acad Radiol. 2014 Sep;21(9):1144-55. doi: 10.1016/j.acra.2014.05.003. Epub 2014 Jul 9. PMID 25022762